CLINICAL TRIAL: NCT01518816
Title: the Role of Serum Total Antioxidant Level in Preterm Labor
Brief Title: Role of Serum Total Antioxidant Level in Preterm Labor
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, Abdallah Salah Abdelatif, THE ROLE OF SERUM TOTAL ANTI OXIDANT IN PRETERM LABOR, Ain Shams Maternity Hospital
Other Study IDs: ABDO-0100
Record Dates: First submitted 2012-01-24; First posted 2012-01-26 (Estimated); Last update posted 2012-01-30 (Estimated); Status verified 2012-01

CONDITIONS: Preterm Labor
Keywords: antioxidant preterm labor
MeSH Terms: conditions — Obstetric Labor, Premature

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: None Retained — serum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- preterm labor cases: Group A: 35 pregnant women diagnosed with preterm labor(Preterm labor pain at least 3 contraction every 20 minutes ,cervical dilatation < 2cm and effacement< 50%) which will deliver within one week maximum after hospitalization.
- control group: Group B: 35 pregnant women( controls )with uncomplicated pregnancies at a similar gestational ages followed routinely in the antenatal care unit.

SUMMARY:
The aim of this study is to detect the association between maternal serum antioxidant level and preterm labor.

DETAILED DESCRIPTION:
Study design:

This is a prospective case-control study.

Setting:

The study will be conducted at Ain Shams University Maternity Hospital.

Population of the study:

A total of 70 pregnant women attending the outpatient obstetric clinic and inpatient of Obstetrics and Gynecology department or when they will be admitted to the delivary room of Ain Shams university hospital.

Patient will be divided in to two groups. Group A: 35 pregnant women diagnosed with preterm labor(Preterm labor pain at least 3 contraction every 20 minutes ,cervical dilatation < 2cm and effacement< 50%) which will deliver within one week maximum after hospitalization.

Group B: 35 pregnant women( controls )with uncomplicated pregnancies at a similar gestational ages followed routinely in the antenatal care unit.

Every case will be subjected to:-

1. Written informed consent before the study.
2. Complete history .
3. Complete general and abdominal examination.
4. Infection markers(CRP,WBCs count, urine analysis ).
5. Gestational age determination by the last menstrual date or Ultrasonography.
6. Local pelvic examination.

ELIGIBILITY:
Inclusion Criteria:

* Preterm labor(pregnant between 28th and 37th week).
* Singleton pregnancy.
* Amnion membranes were intact

Exclusion Criteria:

* Past history of preterm labor or premature delivery.
* Urinary tract infections and any other infections.
* Poly- or oligohydramnios.
* Fetal distress, fetal or uterine anomaly.
* Membranes rupture and placenta pathology.
* Preeclampsia or intrauterine growth retardation

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: pregnant women attending the outpatient obstetric clinic and inpatient of Obstetrics and Gynecology department or when they will be admitted to the delivary room of Ain Shams university hospital.
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2011-10; Primary Completion 2012-04 (Estimated); Study Completion 2012-05 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: ABDALLAH s ABDELATIF, residant, Principal Investigator — Ain Shams Maternity Hospital
Locations (1):
- Ain Shams Maternity Hospital, Cairo, Tertiary, Egypt